CLINICAL TRIAL: NCT02648711
Title: Evaluation of an Alternative Schedule for CRLX101 Alone in Combination With Bevacizumab and in Combination With mFOLFOX6 in Subjects With Advanced Solid Tumor Malignancies
Brief Title: Alternative Dosing for CRLX101(NLG207) Alone, With Avastin and With mFOLFOX6 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRLX101-102
Record Dates: First submitted 2015-11-18; First posted 2016-01-07 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Solid Tumors
Keywords: solid tumors
MeSH Terms: interventions — IT-101; Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRLX101 alone (Experimental): Subjects will receive weekly infusion of CRLX101 alone. Starting dose is 12 mg/m^2 and the next dose level is 15 mg/m^2 (or 10 mg/m^2 if 12 mg/m^2 is not well tolerated. No other dose levels will be explored.
  Interventions: Drug: CRLX101
- CRLX101 in combination with bevacizumab (Experimental): Subjects receive weekly infusion of CRLX101 in combination with bi-weekly bevacizumab (10 mg/kg. The starting dose is 12 mg/m^2 and the next dose level is 15 mg/m^2. No other dose levels will be explored.
  Interventions: Drug: CRLX101; Drug: Bevacizumab
- CRLX101 in combination with mFOLFOX6 (Experimental): Subjects receive weekly infusion of CRLX101 for 3 of every 4 weeks in combination with bi-weekly mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2 and 5FU 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous infusion). The starting dose is 12 mg/m^2 and the next dose level is 15 mg/m^2.
  Interventions: Drug: CRLX101; Drug: mFOLFOX6

INTERVENTIONS:
Drug: CRLX101 — infusion CRLX101 weekly
  Other Names: NLG207
Drug: Bevacizumab — infusion weekly CRLX101 + bevacizumab biweekly
  Other Names: Avastin
  Arms: CRLX101 in combination with bevacizumab
Drug: mFOLFOX6 — infusion weekly CRLX101 for 3 or every 4 weeks and in combination with bi-weekly mFOLFOX6
  Other Names: oxaliplatin, leucovorin, 5FU
  Arms: CRLX101 in combination with mFOLFOX6

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of weekly dosing of CRLX101 (both as monotherapy; (Schedule 1) and in combination with bevacizumab every 2 weeks (Schedule 2) and weekly with a 3 week on / 1 week off schedule in combination with mFOLFOX6 (Schedule 3) to affirm the dose for future clinical studies.

DETAILED DESCRIPTION:
This is an open-label, dose escalation study. Subjects enrolled in Schedule 1 will receive weekly CRLX101 alone. The starting dose for Schedule 1 is 12 mg/m^2 and the next dose level is 15 mg/m^2 (or 10 mg/m^2 if 12 mg/m^2 is not well tolerated). No other dose levels in Schedule 1 will be explored.

Subjects enrolled in Schedule 2 will receive weekly CRLX101 in combination with bi-weekly bevacizumab (10 mg/kg) The starting dose for Schedule 2 is 12 mg/m^ and the next dose is 15 mg/m^2. No other dose levels in Schedule 2 will be explored

Subjects enrolled in Schedule 3 will receive weekly CRLX101 for 3 of every 4 weeks in combination with bi-weekly mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2 and 5FU (fluorouracil) 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous infusion). The starting dose for Schedule 3 is 12 mg/m^2 and the next dose is 15 mg/m^2.

In the absence of dose-limiting toxicities (DLTs) additional subjects may be enrolled (expansion cohort) at the same, intermediate or lower dose levels following consultation between the Investigator and Sponsor.

Enrollment of 6-8 subjects will occur in each cohort for all 3 Schedules.

The MTD is defined as the highest dose level at which fewer than 2 out of 6 subjects experience a DLT. RP2D will be selected based on overall tolerability data from all subjects treated at different dose cohorts in this study.

No intra-patient dose escalation is allowed.

Approximately 61 evaluable subjects are anticipated to be enrolled: 15 subjects in Schedule 1, 15 subjects in Schedule 2 and approximately 31 subjects are anticipated in Schedule 3 (approximately 16 in the dose escalation cohort and up to 15 in the expansion cohort).

The exact number of subjects is dependent on the actual number of subjects enrolled per cohort and the number of cohorts investigated.

ELIGIBILITY:
Inclusion Criteria: (All Subjects)

* Male or female adult subjects ≥18 years of age
* Diagnosis of histologically or cytologically confirmed for:

  * For Schedule 1 and 2: advanced solid tumor malignancy that is refractory to standard therapy and/or for whom no further standard therapy is available
  * For Schedule 3: advanced/metastatic tumors for which mFOLFOX6 is appropriate, or advanced/metastatic tumors that may be sensitive to each component of mFOLFOX6 or sensitive to topoisomerase 1 inhibitors including pancreatic, colorectal, esophageal, gastric, bladder or ovarian cancer, triple-negative breast cancer, small cell lung cancer (SCLC), cholangiocarcinoma, among others
* For Schedules 1 and 2: Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2, For Schedule 3: ECOG Performance Status of 0 or 1
* Life expectancy >12 weeks in the opinion of the Investigator
* Subjects with acceptable pre-study* hematology and biochemistry labs ≤3 days prior to Week 1 Day 1 (W1D1) defined as:

  * absolute neutrophil count (ANC) ≥1.500 cells / µL (1.5 x 10°/L, without growth factor support
  * platelet count ≥100,000 cells/µL (100 x 10° cells/L), without growth factor support
  * hemoglobin ≥9 g/dL (90/g/L)
  * serum total bilirubin ≤1.5 upper limit of normal (ULN), unless Gilbert's disease
  * alanine transaminase (ALT) or aspartate transaminase (AST) ≤2.5 x ULN, (5 x ULN for subjects with liver metastases)
  * calculated or measured creatinine clearance ≥40 mL/min

    * NOTE: If screening hematology and biochemistry labs are performed ≤3 days prior to W1D1, additional pre-study labs do not need to be repeated to confirm eligibility. However, if screening hematology and biochemistry labs are performed greater than 3 days prior to W1D1, additional pre-study labs will need to be performed to confirm continued eligibility to ensure labs remain acceptable per protocol
* Females of childbearing potential must agree to use two effective methods of contraception (or abstain completely from heterosexual intercourse) from the time of informed consent and for 30 days following last dose of study drug

  * NOTE: Females of childbearing potential are defined as women physically capable of becoming pregnant unless the female subject cannot have children due to surgery or other medical reasons (effective tubal ligation, ovaries or the uterus removed, or are post-menopausal). Fertile males of childbearing potential are defined as men who are sexually capable to impregnate the female partner even if surgically sterilized (i.e., vasectomy).

    * highly effective methods of contraception include intra-uterine device (IUD) and hormonal contraception (oral, injectable, patches or implant)
    * effective methods of contraception include barrier methods (latex condom, diaphragm with spermicide, cervical cap, sponge)
    * when possible, subjects should be strongly encouraged to include at least one highly effective method of contraception
* Male subjects must agree to use appropriate method of barrier contraception (latex condom with a spermicidal agent) or abstain completely from heterosexual intercourse fro the time of informed consent and for 120 days following last dose of study drug unless female partner absolutely cannot have children because of surgery or for other medical reasons
* Negative urine pregnancy test
* Ability to understand and willingness to sign a written informed consent form
* Able to comply with study visit schedule and assessments

Exclusion Criteria: (All Subjects)

* Subject has received:

  * chemotherapy or small molecular targeted therapy <2 weeks prior to W1D1
  * approved antibody therapy <5 half-lives from W1D1 (or 4 weeks since last therapy, whichever is the shortest)
  * local palliative radiation <14 days from W1D1
  * invasive surgery requiring general anesthesia <30 days from W1D1
  * chemotherapy with nitrosoureas or mitomycin C <45 days from W1D1
* Uncontrolled grade 2 or greater toxicity except alopecia related to any prior treatment (i.e., chemotherapy, targeted therapy, radiation or surgery) within 7 days prior to W1D1 unless approved by the Medical Monitor
* Prolongation of QT/QTc interval (QTc interval >470) using the Fredericia method of QTc analysis
* Women who are pregnant or nursing
* Any known human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS) or any concurrent infection requiring IV antibiotics
* Any known clinically significant or concurrent acute liver disease, including viral hepatitis
* Primary brain malignant tumors
* Subjects with uncontrolled symptomatic central nervous system (CNS) involvement
* Subjects requiring steroids at stable dose (>4 mg/day dexamethasone or equivalent) for at least 2 weeks
* Uncontrolled hypertension >150/100 mmHg
* Concurrent participation in any other investigational therapeutic study, unless non-interventional study and approved by Sponsor
* History of stroke, deep venous thrombosis (DVT), transient ischemic attack (TIA), unstable angina, or myocardial infarction within 3 months prior to W1D1
* Uncontrolled concurrent disease or illness including but not limited to:

  * symptomatic congestive heart failure (NYHA Class III or IV) per the NYHA Classification, unstable angina pectoris, clinically significant cardiac arrhythmia
  * unstable or untreated cardiac conditions or ejection fraction of <50% as determined by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA)
  * diabetes mellitus (i.e., fasting blood glucose >220 despite acceptable chronic diabetes therapy)
  * psychiatric illness that would limit compliance with study requirements, as determined by the Investigator
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for the study.
* Known hypersensitivity to any component of CRLX101 or excipient or documented medical condition that would prohibit adequate pre-medication with antihistamine.
* Presence of ≥Grade 1 cystitis

Exclusion Criteria for Subjects Enrolled in Schedule 2 Only

* Minor surgical procedure, excluding placement of a vascular access device, within 24 hours prior to W1D1.
* Cardiovascular disease defined as congestive heart failure (NYHA Class II, III, or IV) per the NYHA Classification, angina pectoris requiring nitrate therapy, or myocardial infarction within the last 6 months prior to therapy
* Uncontrolled hypertension (defined as the presence of systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg on two separate occasions. Blood pressure must be controlled to a systolic blood pressure <150 mmHg and/or to diastolic blood pressure <100 mmHg prior to study treatment), or any prior history of hypertensive crisis or hypertensive encephalopathy
* Peripheral vascular disease >Grade 1
* Known congenital long QT syndrome, history of torsades de pointes or ventricular tachycardia.
* Known history of pulmonary hypertension or non-infectious interstitial pneumonitis.
* History or evidence of thrombotic or hemorrhagic disorders: including cerebrovascular accident (CVA) / stroke or transient ischemic attack (TIA), intracerebral hemorrhage or sub- arachnoid hemorrhage ≤ 6 months prior to W1D1
* Chronic daily aspirin >325 mg/day or clopidogrel (>75 mg/day)
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization
* Any of the following serious, non-healing conditions:wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either: urine dipstick ≥2+ (subjects discovered to have a ≥2+ proteinuria on dipstick urinalysis at baseline should undergo 24-hour urine collection and must demonstrate <1g of protein in 24 hours to be eligible): 24-hour urine collection demonstrates >1g of protein in 24 hours
* Immunocompromised subjects, including known seropositivity for human immunodeficiency virus (HIV), or current or chronic hepatitis B and/or hepatitis C infection (as detected by positive testing for hepatitis B surface antigen [HbsAg] or antibody to hepatitis C virus [anti HCV] with confirmatory testing). [Note: testing is not mandatory to be eligible for the study. However, if a subject is at risk for having undiagnosed hepatitis C virus (HCV) (due to history of injection drug use or due to geographic location for example), testing at screening should be considered]
* Chronic treatment with corticosteroids (prednisone >12.5 mg/day or dexamethasone >2 mg/day excluding inhaled steroids

Exclusion Criteria for Subjects Enrolled in Schedule 3 Only

* Known hypersensitivity to 5FU, oxaliplatin or other platinum agent, or to their excipients
* Known dihydropyridine dehydrogenase (DPD) enzyme deficiency (testing not required)
* Baseline peripheral neuropathy grade ≥ 2
* Progressive disease within ≤ 6 months of completing an oxaliplatin containing adjuvant therapy
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10-17 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD), Recommended Phase 2 Dose (RP2D) | 15 months
  To determine the maximum tolerated dose (MTD) / recommended Phase 2 dose (RP2D) of CRLX101 when administered by intravenous (IV) infusion every week (QW) alone (Schedule 1), (QW) in combination with bevacizumab (Q2W) (Schedule 2) and weekly with a 3-week on / 1-week off schedule in combination with mFOLFOX6 (Q2W) (Schedule 3) in subjects with advanced solid tumor malignancies

SECONDARY OUTCOMES:
Safety and Tolerability (Weekly Dosing) determined by reported adverse events, serious adverse events, physical exam findings, vital sign measurements,12-lead ECG readings, clinical lab evaluations, and treatment discontinuation due to toxicity. | 15 months
  Will be determined by reported AEs, SAEs, physical exam findings, vital sign measurements,12-lead ECG readings, clinical lab evaluations, and treatment discontinuation due to toxicity.
Pharmacokinetic Profile (PK) - Urine | 15 months
  Urine samples will be collected to evaluate the urinary excretion of total and unconjugated drug before, during, and after infusion. PK parameters in urine will include the maximum concentration (Cmax), amount of drug in the urine, % of drug eliminated in the urine. PK parameters will be calculated using non-compartmental analysis. Actual sampling times will be used to calculate PK parameters in this study.
Pharmacokinetic Profile (PK) - Plasma:CL | 15 months
  Plasma PK parameters will include clearance (CL) for both total and unconjugated drug.
Pharmacokinetic Profile (PK) - Plasma:Vd | 15 months
  The plasma PK parameters will include volume of distribution (Vd)
Pharmacokinetic Profile (PK) - Plasma:t1/2 | 15 months
  Plasma PK parameters will include half-life (t1/2)
Pharmacokinetic Profile (PK) - Plasma:Cmax | 15 months
  Plasma PK parameters will include maximum concentration (Cmax)
Pharmacokinetic Profile (PK) - Plasma:AUC | 15 months
  Plasma PK parameters will include area under the concentration versus time curve (AUC)
Anti-tumor Activity | 15 months
  To further explore preliminary signs of anti-tumor activity of CRLX101 when administered alone (Schedule 1) and in combination with bevacizumab (Schedule 2), and in combination with mFOLFOX6 (Schedule 3)

CONTACTS AND LOCATIONS:
Overall Officials: NewLink Ge, Study Chair — NewLink Genetics Inc
Locations (3):
- United States (3):
  - START Midwest/Cancer & Hematology Centers of Western Michigan, PC, Grand Rapids, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kummar S, Raffeld M, Juwara L, Horneffer Y, Strassberger A, Allen D, Steinberg SM, Rapisarda A, Spencer SD, Figg WD, Chen X, Turkbey IB, Choyke P, Murgo AJ, Doroshow JH, Melillo G. Multihistology, target-driven pilot trial of oral topotecan as an inhibitor of hypoxia-inducible factor-1alpha in advanced solid tumors. Clin Cancer Res. 2011 Aug 1;17(15):5123-31. doi: 10.1158/1078-0432.CCR-11-0682. Epub 2011 Jun 14. PMID 21673063
- [Background] Eliasof S, Lazarus D, Peters CG, Case RI, Cole RO, Hwang J, Schluep T, Chao J, Lin J, Yen Y, Han H, Wiley DT, Zuckerman JE, Davis ME. Correlating preclinical animal studies and human clinical trials of a multifunctional, polymeric nanoparticle. Proc Natl Acad Sci U S A. 2013 Sep 10;110(37):15127-32. doi: 10.1073/pnas.1309566110. Epub 2013 Aug 26. PMID 23980155
- [Background] Schluep T, Hwang J, Cheng J, Heidel JD, Bartlett DW, Hollister B, Davis ME. Preclinical efficacy of the camptothecin-polymer conjugate IT-101 in multiple cancer models. Clin Cancer Res. 2006 Mar 1;12(5):1606-14. doi: 10.1158/1078-0432.CCR-05-1566. PMID 16533788
- [Background] Numbenjapon T, Wang J, Colcher D, Schluep T, Davis ME, Duringer J, Kretzner L, Yen Y, Forman SJ, Raubitschek A. Preclinical results of camptothecin-polymer conjugate (IT-101) in multiple human lymphoma xenograft models. Clin Cancer Res. 2009 Jul 1;15(13):4365-73. doi: 10.1158/1078-0432.CCR-08-2619. Epub 2009 Jun 23. PMID 19549776
- [Background] Pham E, Birrer MJ, Eliasof S, Garmey EG, Lazarus D, Lee CR, Man S, Matulonis UA, Peters CG, Xu P, Krasner C, Kerbel RS. Translational impact of nanoparticle-drug conjugate CRLX101 with or without bevacizumab in advanced ovarian cancer. Clin Cancer Res. 2015 Feb 15;21(4):808-18. doi: 10.1158/1078-0432.CCR-14-2810. Epub 2014 Dec 18. PMID 25524310
- [Background] Gaur S, Chen L, Yen T, Wang Y, Zhou B, Davis M, Yen Y. Preclinical study of the cyclodextrin-polymer conjugate of camptothecin CRLX101 for the treatment of gastric cancer. Nanomedicine. 2012 Jul;8(5):721-30. doi: 10.1016/j.nano.2011.09.007. Epub 2011 Oct 25. PMID 22033079
- [Background] Rapisarda A, Melillo G. Overcoming disappointing results with antiangiogenic therapy by targeting hypoxia. Nat Rev Clin Oncol. 2012 Apr 24;9(7):378-90. doi: 10.1038/nrclinonc.2012.64. PMID 22525710
- [Background] Rapisarda A, Zalek J, Hollingshead M, Braunschweig T, Uranchimeg B, Bonomi CA, Borgel SD, Carter JP, Hewitt SM, Shoemaker RH, Melillo G. Schedule-dependent inhibition of hypoxia-inducible factor-1alpha protein accumulation, angiogenesis, and tumor growth by topotecan in U251-HRE glioblastoma xenografts. Cancer Res. 2004 Oct 1;64(19):6845-8. doi: 10.1158/0008-5472.CAN-04-2116. PMID 15466170
- [Background] Conley SJ, Baker TL, Burnett JP, Theisen RL, Lazarus D, Peters CG, Clouthier SG, Eliasof S, Wicha MS. CRLX101, an investigational camptothecin-containing nanoparticle-drug conjugate, targets cancer stem cells and impedes resistance to antiangiogenic therapy in mouse models of breast cancer. Breast Cancer Res Treat. 2015 Apr;150(3):559-67. doi: 10.1007/s10549-015-3349-8. Epub 2015 Apr 2. PMID 25833208
- [Background] Escudier B, Pluzanska A, Koralewski P, Ravaud A, Bracarda S, Szczylik C, Chevreau C, Filipek M, Melichar B, Bajetta E, Gorbunova V, Bay JO, Bodrogi I, Jagiello-Gruszfeld A, Moore N; AVOREN Trial investigators. Bevacizumab plus interferon alfa-2a for treatment of metastatic renal cell carcinoma: a randomised, double-blind phase III trial. Lancet. 2007 Dec 22;370(9605):2103-11. doi: 10.1016/S0140-6736(07)61904-7. PMID 18156031
- [Background] Weiss GJ, Chao J, Neidhart JD, Ramanathan RK, Bassett D, Neidhart JA, Choi CHJ, Chow W, Chung V, Forman SJ, Garmey E, Hwang J, Kalinoski DL, Koczywas M, Longmate J, Melton RJ, Morgan R, Oliver J, Peterkin JJ, Ryan JL, Schluep T, Synold TW, Twardowski P, Davis ME, Yen Y. First-in-human phase 1/2a trial of CRLX101, a cyclodextrin-containing polymer-camptothecin nanopharmaceutical in patients with advanced solid tumor malignancies. Invest New Drugs. 2013 Aug;31(4):986-1000. doi: 10.1007/s10637-012-9921-8. Epub 2013 Feb 9. PMID 23397498
- [Background] Griggs JJ, Mangu PB, Anderson H, Balaban EP, Dignam JJ, Hryniuk WM, Morrison VA, Pini TM, Runowicz CD, Rosner GL, Shayne M, Sparreboom A, Sucheston LE, Lyman GH; American Society of Clinical Oncology. Appropriate chemotherapy dosing for obese adult patients with cancer: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2012 May 1;30(13):1553-61. doi: 10.1200/JCO.2011.39.9436. Epub 2012 Apr 2. PMID 22473167
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Keefe, SM, Heitjan D, Hennessy M., et al. Interim results of a phase 1b/2a study evaluating the nano pharmaceutical CRLX101 with bevacizumab (bev) in the treatment of subjects (pts) with refractory metastatic renal cell carcinoma (mRCC). J Clin Oncol 32, 2014 (suppl 4; abstr 412).
- [Background] Yen et al, Final phase 1/2a results evaluating the cyclodextrin-containing nanoparticle CRLX101 in subjects with advanced solid tumor malignancies, 23rd EORTC-NCI-AACR, Nov 12-16, 2011: abstract A97
- [Background] Guichard S, Arnould S, Hennebelle I, Bugat R, Canal P. Combination of oxaliplatin and irinotecan on human colon cancer cell lines: activity in vitro and in vivo. Anticancer Drugs. 2001 Oct;12(9):741-51. doi: 10.1097/00001813-200110000-00006. PMID 11593056
- [Background] Zeghari-Squalli N, Raymond E, Cvitkovic E, Goldwasser F. Cellular pharmacology of the combination of the DNA topoisomerase I inhibitor SN-38 and the diaminocyclohexane platinum derivative oxaliplatin. Clin Cancer Res. 1999 May;5(5):1189-96. PMID 10353756
- [Background] Bissery MC, Vrignaud P, Lavelle F. In vivo evaluation of the irinotecan-oxaliplatin combination. Proc Am Assoc Cancer Res 1998; 39: 526.
- [Background] Goldwasser F, Bozec L, Zeghari-Squalli N, Misset JL. Cellular pharmacology of the combination of oxaliplatin with topotecan in the IGROV-1 human ovarian cancer cell line. Anticancer Drugs. 1999 Feb;10(2):195-201. doi: 10.1097/00001813-199902000-00008. PMID 10211550
- [Background] Ychou M, Conroy T, Seitz JF, Gourgou S, Hua A, Mery-Mignard D, Kramar A. An open phase I study assessing the feasibility of the triple combination: oxaliplatin plus irinotecan plus leucovorin/ 5-fluorouracil every 2 weeks in patients with advanced solid tumors. Ann Oncol. 2003 Mar;14(3):481-9. doi: 10.1093/annonc/mdg119. PMID 12598357
- [Background] Lee J, Kang WK, Kwon JM, Oh SY, Lee HR, Kim HJ, Park BB, Lim HY, Han MJ, Park JO, Park YS. Phase II trial of irinotecan plus oxaliplatin and 5-fluorouracil/leucovorin in patients with untreated metastatic gastric adenocarcinoma. Ann Oncol. 2007 Jan;18(1):88-92. doi: 10.1093/annonc/mdl317. Epub 2006 Sep 13. PMID 16971670
- [Background] Long HJ 3rd, Bundy BN, Grendys EC Jr, Benda JA, McMeekin DS, Sorosky J, Miller DS, Eaton LA, Fiorica JV; Gynecologic Oncology Group Study. Randomized phase III trial of cisplatin with or without topotecan in carcinoma of the uterine cervix: a Gynecologic Oncology Group Study. J Clin Oncol. 2005 Jul 20;23(21):4626-33. doi: 10.1200/JCO.2005.10.021. Epub 2005 May 23. PMID 15911865
- [Background] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Background] Souglakos J, Androulakis N, Syrigos K, Polyzos A, Ziras N, Athanasiadis A, Kakolyris S, Tsousis S, Kouroussis Ch, Vamvakas L, Kalykaki A, Samonis G, Mavroudis D, Georgoulias V. FOLFOXIRI (folinic acid, 5-fluorouracil, oxaliplatin and irinotecan) vs FOLFIRI (folinic acid, 5-fluorouracil and irinotecan) as first-line treatment in metastatic colorectal cancer (MCC): a multicentre randomised phase III trial from the Hellenic Oncology Research Group (HORG). Br J Cancer. 2006 Mar 27;94(6):798-805. doi: 10.1038/sj.bjc.6603011. PMID 16508637
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] Assenat E, Desseigne F, Thezenas S, Viret F, Mineur L, Kramar A, Samalin E, Portales F, Bibeau F, Crapez-Lopez E, Bleuse JP, Ychou M. Cetuximab plus FOLFIRINOX (ERBIRINOX) as first-line treatment for unresectable metastatic colorectal cancer: a phase II trial. Oncologist. 2011;16(11):1557-64. doi: 10.1634/theoncologist.2011-0141. Epub 2011 Oct 20. PMID 22016477
- [Background] Conroy T, Paillot B, Francois E, Bugat R, Jacob JH, Stein U, Nasca S, Metges JP, Rixe O, Michel P, Magherini E, Hua A, Deplanque G. Irinotecan plus oxaliplatin and leucovorin-modulated fluorouracil in advanced pancreatic cancer--a Groupe Tumeurs Digestives of the Federation Nationale des Centres de Lutte Contre le Cancer study. J Clin Oncol. 2005 Feb 20;23(6):1228-36. doi: 10.1200/JCO.2005.06.050. PMID 15718320
- [Background] Ychou M, Desseigne F, Guimbaud R et al. Randomized phase II trial comparing folfirinox (5FU/leucovorin [LV], irinotecan [I] and oxaliplatin [O] vs gemcitabine (G) as first-line treatment for metastatic pancreatic adenocarcinoma (MPA). First results of the ACCORD 11 trial [abstract]. J Clin Oncol 2007;25(June 20 Suppl):4516.
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Cremolini C, Loupakis F, Antoniotti C, Lupi C, Sensi E, Lonardi S, Mezi S, Tomasello G, Ronzoni M, Zaniboni A, Tonini G, Carlomagno C, Allegrini G, Chiara S, D'Amico M, Granetto C, Cazzaniga M, Boni L, Fontanini G, Falcone A. FOLFOXIRI plus bevacizumab versus FOLFIRI plus bevacizumab as first-line treatment of patients with metastatic colorectal cancer: updated overall survival and molecular subgroup analyses of the open-label, phase 3 TRIBE study. Lancet Oncol. 2015 Oct;16(13):1306-15. doi: 10.1016/S1470-2045(15)00122-9. Epub 2015 Aug 31. PMID 26338525
- [Background] Marsh Rde W, Talamonti MS, Katz MH, Herman JM. Pancreatic cancer and FOLFIRINOX: a new era and new questions. Cancer Med. 2015 Jun;4(6):853-63. doi: 10.1002/cam4.433. Epub 2015 Feb 19. PMID 25693729
- [Background] Lowery MA, Yu KH, Adel NG et al. Activity of front-line FOLFIRINOX (FFX) in stage III/IV pancreatic adenocarcinoma (PC) at Memorial Sloan-Kettering Cancer Center (MSKCC) [abstract]. ASCO Meeting Abstracts 2012;30:4057.
- [Background] Clark AJ, Wiley DT, Zuckerman JE, Webster P, Chao J, Lin J, Yen Y, Davis ME. CRLX101 nanoparticles localize in human tumors and not in adjacent, nonneoplastic tissue after intravenous dosing. Proc Natl Acad Sci U S A. 2016 Apr 5;113(14):3850-4. doi: 10.1073/pnas.1603018113. Epub 2016 Mar 21. PMID 27001839
- [Background] Castells MC, Tennant NM, Sloane DE, Hsu FI, Barrett NA, Hong DI, Laidlaw TM, Legere HJ, Nallamshetty SN, Palis RI, Rao JJ, Berlin ST, Campos SM, Matulonis UA. Hypersensitivity reactions to chemotherapy: outcomes and safety of rapid desensitization in 413 cases. J Allergy Clin Immunol. 2008 Sep;122(3):574-80. doi: 10.1016/j.jaci.2008.02.044. Epub 2008 May 27. PMID 18502492
- [Background] Leong S, Eckhardt SG, Chan E, Messersmith WA, Spratlin J, Camidge DR, Diab S, Khosravan R, Lin X, Chow Maneval E, Lockhart AC. A phase I study of sunitinib combined with modified FOLFOX6 in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2012 Jul;70(1):65-74. doi: 10.1007/s00280-012-1880-4. Epub 2012 May 24. PMID 22623210
- [Background] Smith TJ, Bohlke K, Lyman GH, Carson KR, Crawford J, Cross SJ, Goldberg JM, Khatcheressian JL, Leighl NB, Perkins CL, Somlo G, Wade JL, Wozniak AJ, Armitage JO; American Society of Clinical Oncology. Recommendations for the Use of WBC Growth Factors: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2015 Oct 1;33(28):3199-212. doi: 10.1200/JCO.2015.62.3488. Epub 2015 Jul 13. PMID 26169616
- [Background] Sriram D, Yogeeswari P, Thirumurugan R, Bal TR. Camptothecin and its analogues: a review on their chemotherapeutic potential. Nat Prod Res. 2005 Jun;19(4):393-412. doi: 10.1080/14786410412331299005. PMID 15938148
- [Background] Rouch JA, Burton B, Dabb A, Brown V, Seung AH, Kinsman K, Holdhoff M. Comparison of enteral and parenteral methods of urine alkalinization in patients receiving high-dose methotrexate. J Oncol Pharm Pract. 2017 Jan;23(1):3-9. doi: 10.1177/1078155215610914. Epub 2016 Jun 23. PMID 26467268
- [Background] Sharma S, Abhyankar V, Burgess RE, Infante J, Trowbridge RC, Tarazi J, Kim S, Tortorici M, Chen Y, Robles RL. A phase I study of axitinib (AG-013736) in combination with bevacizumab plus chemotherapy or chemotherapy alone in patients with metastatic colorectal cancer and other solid tumors. Ann Oncol. 2010 Feb;21(2):297-304. doi: 10.1093/annonc/mdp489. Epub 2009 Nov 25. PMID 19940012